CLINICAL TRIAL: NCT01921335
Title: Phase I Dose-escalation Trial of ARRY-380 in Combination With Trastuzumab in Participants With Brain Metastases From HER2+ Breast Cancer
Brief Title: ARRY-380 + Trastuzuamab for Breast w/ Brain Mets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Array BioPharma (Industry); Breast Cancer Research Foundation (Other)
Responsible Party: Principal Investigator, Nancy Lin, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-198; ARRAY-380-104X (Other Grant/Funding Number: Array BioPharma)
Record Dates: First submitted 2013-08-02; First posted 2013-08-13 (Estimated); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Brain Metastases From HER2 and Breast Cancer; Advanced HER2-positive Breast Cancer
Keywords: ARRY-380; Trastuzumab; Advanced HER2-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ARRY-380 Twice Daily Dosage (Active Comparator): ARRY-380 will be 450mg orally twice-daily. Trastuzumab will be given at the standard full dose with a loading dose of 8 mg/kg on Day 1, cycle 1, followed by 6 mg/kg in subsequent cycles. Participants who are within 5 weeks of a 6 mg/kg dose or within 2 weeks of a 2 mg/kg dose of trastuzumab at the time of initial study dosing will not be required to have a re-loading dose but will begin treatment at 6 mg/kg.ARRY-380 will be escalated until MTD is defined or the maximum planned dose has been evaluated. The dose for subsequent dose levels will be determined according to the treatment-related AE observed during the cycle 1 (21 days) in the previous dose level
  Interventions: Drug: ARRY-380 Twice Daily Dosage; Drug: Trastuzumab
- ARRY-380 Once Daily (Active Comparator): ARRY-380 will be 750mg orally once-daily. Trastuzumab will be given at the standard full dose with a loading dose of 8 mg/kg on Day 1, cycle 1, followed by 6 mg/kg in subsequent cycles. Participants who are within 5 weeks of a 6 mg/kg dose or within 2 weeks of a 2 mg/kg dose of trastuzumab at the time of initial study dosing will not be required to have a re-loading dose but will begin treatment at 6 mg/kg. ARRY-380 will be escalated until MTD is defined or the maximum planned dose has been evaluated. The dose for subsequent dose levels will be determined according to the treatment-related AE observed during the cycle 1 (21 days) in the previous dose level
  Interventions: Drug: ARRY-380 Once Daily; Drug: Trastuzumab

INTERVENTIONS:
Drug: ARRY-380 Twice Daily Dosage — ARRY-380 will be administered daily (either twice-daily along with concurrent administration of trastuzumab on Day 1. PK sampling of ARRY-380 is planned on Day 15. Blood samples will be collected at pre-dosing, 2 hours (± 1 hour), and 6 hours (± 2 hours). The same time points will be collected for BID and QD schedules. On the PK collection day participants should fast one hour before and one hour after taking ARRY-380.
  Arms: ARRY-380 Twice Daily Dosage
Drug: ARRY-380 Once Daily — ARRY-380 will be administered daily once-daily) along with concurrent administration of trastuzumab on Day 1. PK sampling of ARRY-380 is planned on Day 15. Blood samples will be collected at pre-dosing, 2 hours (± 1 hour), and 6 hours (± 2 hours). The same time points will be collected for BID and QD schedules. On the PK collection day participants should fast one hour before and one hour after taking ARRY-380.
  Arms: ARRY-380 Once Daily
Drug: Trastuzumab — 6 mg/kg IV every 3 weeks
  Other Names: Herceptin

SUMMARY:
The purpose of this study is to test the safety of different doses of ARRY-380 in combination with trastuzumab. Trastuzumab is an FDA approved drug for the treatment of HER2 metastatic breast cancer. However, the combination of ARRY-380 and trastuzumab has not yet been tested. Both agents block the HER2 receptor, which is thought to be overactive in HER2-positive breast cancer. It is thought that ARRY-380 and trastuzumab might work together because they attach to different parts of the HER2 receptor and prevent it from functioning. Because HER2 positive breast cancer contains high levels of HER2 receptor, but normal cells in your body generally do not, the drugs may be able to "target" the cancer cells. In addition, in laboratory studies, ARRY-380 appears to have some penetration into the brain.

DETAILED DESCRIPTION:
If a patient participates in this research study, the patient will receive ARRY-380 and a drug-dosing diary to record when the patient took ARRY-380 for each study treatment cycle. Each study treatment cycle will last for 3 weeks (21 days) during which time the patient will be taking ARRY-380 by mouth every day. At the time the patient enters the study, the patient will be assigned to either Arm A or Arm B. The difference between the two study arms includes ARRY-380 administered twice-daily (morning and evenings - Arm A) or once-daily (morning - Arm B). The patient will also be given Trastuzumab by intravenous infusion (by vein) on day 1 of each cycle (same dose and schedule for both study arms).

The dose of trastuzumab will be the same for everyone on study, and will be the standard approved dose for this medication. In the first portion of the study, the investigators will examine the effects of different dose of ARRY-380 when given in combination with trastuzumab. Initially, 3 participants will be treated with a low dose of the ARRY-380 in combination with standard dose of trastuzumab. If this dose does not cause intolerable side effects, more participants may receive the drug combination at the same dose. The patient will be informed of the assigned dose when the patient enters the study. The patient will be asked to take ARRY-380 for as long as the study treatment is of possible benefit to the patient. After the patient is finished taking ARRY-380, the study doctor will ask the patient to visit the office for follow-up exams for at least one more visit within 4 weeks of the patient's last study treatment.

At the start of each cycle the patient will have:

* A medical history, which includes questions about health, current medications, and any allergies.
* Performance status, which evaluates the ability to carry on with usual activities.
* Physical examination, the doctor will examine the patient body, including measuring height, weight, and vital signs (blood pressure, body temperature, pulse rate and breathing rate).
* A neurological examination to asses any neurological symptoms(for example, difficulties with balance)
* Blood tests will be drawn at the beginning of each study treatment cycle for tests to monitor the function of liver and kidneys and to check blood cell counts. In addition, blood tests will be drawn on days 4, 8, and 15 of the first cycle of study treatment to monitor liver function.

Periodically the patient will undergo:

* The patient will have a brain MRI every two cycles. If the brain scans are stable or improved after the patient has been on the study for 6 months or longer, the frequency of your body scans will be decreased to once every 4 cycles. The patient will also have CT or MRI scans of the body at the end of cycle 2, cycle 4 and every 4 cycles thereafter. The research doctor may ask the patient to have a bone scan at the same time points if this is clinically indicated.
* Electrocardiogram (EKG), which shows the electrical activity of the heart. It will be performed on Day 1 of cycle 2.
* Echocardiogram (ECHO) (ultrasound of the heart) or MUGA scan (test of heart function using a small amount of a radioactive substance). This will be performed every 3-4 months.

Additional research procedures to be performed:

* On Cycle 1, Day 15 blood for ("PK") pharmacokinetic (what the body does to the drug) sampling will be drawn before the morning dose of ARRY-380, after 2 hours and after six hours.
* Blood tests for research, which will include about 2 tablespoons of blood collected before cycle 1 and after coming off study treatment. In general terms, scientists will study the genes, the RNA, and the proteins that are found in the blood samples. Scientists will also measure and characterize circulating tumor cells in the blood, if they are present. In addition, these specimens may be tested with new types of tests, as they become available. Results of the research tests on blood will not be reported back to the patient.
* Archival Tumor Tissue Sample: A sample (or samples) of the patient's tumor tissue (from a past surgery and/or biopsy) will be collected and used to learn more about the development of metastatic breast cancer. In general terms, scientists will study the genes, the RNA, and the proteins that are found both in breast tumors and in normal tissue. In addition, these specimens may be tested with new types of tests, as they become available. Laboratory-based investigators conducting this research will not have access to patient identification information such as name or medical record number. Results of the research tests on tissue will not be reported back to the patient.

After the final dose of the study drug:

The patient will have a follow-up visit one month after coming off study treatment. During that visit, the patient will have a physical examination, functional assessment, assessment of any toxicities and current medications. If the patient continues to have ongoing side effects related to the study treatment, the investigators will continue to follow the patient until these side effects resolve. If the patient withdrew from the study for another reason other than tumor progression, the patient will continue to be followed until tumor progression.

Planned Follow-up:

The investigators would like to keep track of the patient's medical condition indefinitely. The investigators would like to do this either by seeing the patient in clinic or by contacting the patient and the patient's primary doctor periodically to see how the patient is doing. Keeping in touch with the patient and checking the patient's condition periodically helps the investigators look at the long-term effects of the research study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the following criteria on screening examination to be eligible to participate in the study. Laboratory evaluations must have been performed within 14 days of study entry. Non-laboratory tests must have been performed within 30 days of study entry. Evaluation of LVEF must have been performed within 60 days of study entry:
* Participants must have histologically confirmed HER2+ (3+ by immunohistochemistry and/or FISH ratio >/= 2.0) invasive breast cancer. Central confirmation of HER2 status is not required.
* Participants must have measurable CNS disease, defined as at least one parenchymal brain lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 10 mm by local radiology review (note: measurable non-CNS disease is NOT required for study participation). See section 10 for the evaluation of measureable disease.
* New or progressive CNS lesions, as assessed by the patient's treating physician.
* It is anticipated that some participants may have multiple progressive CNS lesions, one or several of which are treated with SRS or surgery with residual un-treated lesions remaining. Such participants are eligible for enrollment on this study providing that at least one untreated lesion is measurable, as defined in section 3.1.2. The location of the measurable lesion should be documented in the patient chart and case report form.
* Participants who have had prior cranial surgery are eligible, provided that there is evidence of measurable residual or progressive lesions. If a patient has surgical resection followed by WBRT, then there must be evidence of progressive CNS disease after the completion of WBRT.
* Participants who have had prior WBRT and/or SRS and then whose lesions have progressed thereafter are also eligible. In this case, lesions which have been treated with SRS may be considered as target lesions if there is unequivocal evidence, in the opinion of the treating physician, of progression following SRS.
* Participants who have not previously been treated with cranial radiation (e.g. WBRT or SRS) are eligible to enter the study, but such participants must be asymptomatic from their CNS metastases and not requiring corticosteroids.
* No increase in corticosteroid dose in the week prior to the baseline brain MRI.
* Age ≥18 years
* ECOG performance status 0 to 2 (see Appendix A)
* Participants must have normal organ and marrow function as defined below:
* Absolute neutrophil count ≥ 1,000/mcL
* Platelets ≥ 75,000/mcL
* Total bilirubin < 2 X institutional upper limit of normal
* AST (SGOT)/ALT (SGPT) < 2.5 X institutional upper limit of normal in participants without liver metastases and < 5 ULN in participants with documented liver metastases
* Left ventricular ejection fraction ≥ 50%, as determined by RVG or echocardiogram within 60 days prior to initiation of protocol therapy
* Prior therapy - Prior trastuzumab and/or lapatinib are allowed. There is no limit on the number of prior lines of therapy.
* The effects of ARRY-380 on the developing human fetus are unknown. For this reason and because other therapeutic agents used in this trial may be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study.
* Participants who have had chemotherapy or radiotherapy within 14 days prior to entering the study (with the exception of trastuzumab) or those who have not recovered from adverse events to ≤ grade 1 due to agents administered more than 4 weeks earlier.
* Participants may not be receiving any other investigational agents. Concurrent treatment with bisphosphonates or denosumab is allowed
* History of grade 3 or 4 allergic reactions attributed to compounds of similar chemical or biologic composition to ARRY-380 or trastuzumab
* Known contraindication to MRI with gadolinium contrast, such as cardiac pacemaker, shrapnel, or ocular foreign body
* Leptomeningeal carcinomatosis as the only site of CNS involvement
* More than 2 seizures over the last 4 weeks prior to study entry
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnancy (positive pregnancy test) or lactation
* Individuals with a history of a different active malignancy are ineligible. Participants with a history of other malignancies are eligible if they have been disease-free for at least 2 years, not on active treatment, and deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 2 years: cervical cancer in situ, basal cell or squamous cell carcinoma of the skin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Determine Maximum-tolerated dose of ARRY-380 with Trastuzumab | 2 years
  To determine the maximum-tolerated dose (MTD) and recommended phase 2 dose (RP2D) of ARRY-380 in combination with trastuzumab in participants with HER2+ breast cancer and central nervous system (CNS metastasis)

SECONDARY OUTCOMES:
CNS objective response rate according to volumetric criteria | 2 Years
  CNS objective response rate according to volumetric criteria
Non-CNS objective response rate according to RECIST 1.1 | 2 years
  Non-CNS objective response rate according to RECIST 1.1
Proportion of participants with stable or responsive disease in both CNS and non-CNS at 16 and 24 weeks. | 2 Years
  Proportion of participants with stable or responsive disease in both CNS and non-CNS at 16 and 24 weeks.
Progression-free survival | 2 Years
  Progression-free survival
Clinical benefit (CR, PR, or SD>/=24 weeks) | 2 Years
  Clinical benefit (CR, PR, or SD>/=24 weeks)
Overall survival | 2 Years
  Overall survival
CNS Response according to modified RECIST 1.1 | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Lin, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Metzger Filho O, Leone JP, Li T, Tan-Wasielewski Z, Trippa L, Barry WT, Younger J, Lawler E, Walker L, Freedman RA, Tolaney SM, Krop I, Winer EP, Lin NU. Phase I dose-escalation trial of tucatinib in combination with trastuzumab in patients with HER2-positive breast cancer brain metastases. Ann Oncol. 2020 Sep;31(9):1231-1239. doi: 10.1016/j.annonc.2020.05.014. Epub 2020 May 24. PMID 32461105